CLINICAL TRIAL: NCT03860857
Title: The BEACoN Study- Biomarker Exploration in Aging, Cognition and Neurodegeneration
Brief Title: Biomarker Exploration in Aging, Cognition and Neurodegeneration
Acronym: BEACoN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Michael Yassa, Professor, University of California, Irvine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20173832; R01AG053555 (NIH)
Record Dates: First submitted 2019-02-15; First posted 2019-03-04 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer Disease; Cognitive Impairment; Cognitive Decline
Keywords: Alzheimer disease; cognitive impairment; mild cognitive impairment; biomarker; MRI; PET
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: All participants will complete the same study procedures, including the tau PET scans with investigational radio tracer 18F-MK6240. The arms define the age range and APOE status of the participants, with each having their own enrollment target.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Age 60-65 ApoE e4+ (Experimental): Participants in this cohort are between the ages of 60-65 and are ApoE e4 carriers. All participants in this cohort will complete the Amyloid PET scan, Tau PET scan using MK-6240, MRI scans, and neurocognitive testing.
  Interventions: Radiation: Amyloid PET scan; Drug: Tau PET scan using MK-6240; Behavioral: Neurocognitive testing; Other: MRI
- Age 66-70 ApoE e4- (Experimental): Participants in this cohort are between the ages of 66-70 and are not ApoE e4 carriers. All participants in this cohort will complete the Amyloid PET scan, Tau PET scan using MK-6240, MRI scans, and neurocognitive testing.
  Interventions: Radiation: Amyloid PET scan; Drug: Tau PET scan using MK-6240; Behavioral: Neurocognitive testing; Other: MRI
- Age 66-70 ApoE e4+ (Experimental): Participants in this cohort are between the ages of 66-70 and are ApoE e4 carriers. All participants in this cohort will complete the Amyloid PET scan, Tau PET scan using MK-6240, MRI scans, and neurocognitive testing.
  Interventions: Radiation: Amyloid PET scan; Drug: Tau PET scan using MK-6240; Behavioral: Neurocognitive testing; Other: MRI
- Age 71-75 ApoE e4- (Experimental): Participants in this cohort are between the ages of 71-75 and are not ApoE e4 carriers. All participants in this cohort will complete the Amyloid PET scan, Tau PET scan using MK-6240, MRI scans, and neurocognitive testing.
  Interventions: Radiation: Amyloid PET scan; Drug: Tau PET scan using MK-6240; Behavioral: Neurocognitive testing; Other: MRI
- Age 71-75 ApoE e4+ (Experimental): Participants in this cohort are between the ages of 71-75 and are ApoE e4 carriers. All participants in this cohort will complete the Amyloid PET scan, Tau PET scan using MK-6240, MRI scans, and neurocognitive testing.
  Interventions: Radiation: Amyloid PET scan; Drug: Tau PET scan using MK-6240; Behavioral: Neurocognitive testing; Other: MRI
- Age 76-80 ApoE e4- (Experimental): Participants in this cohort are between the ages of 76-80 and are not ApoE e4 carriers. All participants in this cohort will complete the Amyloid PET scan, Tau PET scan using MK-6240, MRI scans, and neurocognitive testing.
  Interventions: Radiation: Amyloid PET scan; Drug: Tau PET scan using MK-6240; Behavioral: Neurocognitive testing; Other: MRI
- Age 76-80 ApoE e4+ (Experimental): Participants in this cohort are between the ages of 76-80 and are ApoE e4 carriers. All participants in this cohort will complete the Amyloid PET scan, Tau PET scan using MK-6240, MRI scans, and neurocognitive testing.
  Interventions: Radiation: Amyloid PET scan; Drug: Tau PET scan using MK-6240; Behavioral: Neurocognitive testing; Other: MRI
- Age 81+ ApoE e4- (Experimental): Participants in this cohort are between the ages of 81-85 and are not ApoE e4 carriers. All participants in this cohort will complete the Amyloid PET scan, Tau PET scan using MK-6240, MRI scans, and neurocognitive testing.
  Interventions: Radiation: Amyloid PET scan; Drug: Tau PET scan using MK-6240; Behavioral: Neurocognitive testing; Other: MRI
- Age 81+ ApoE e4+ (Experimental): Participants in this cohort are between the ages of 81-85 and are ApoE e4 carriers. All participants in this cohort will complete the Amyloid PET scan, Tau PET scan using MK-6240, MRI scans, and neurocognitive testing.
  Interventions: Radiation: Amyloid PET scan; Drug: Tau PET scan using MK-6240; Behavioral: Neurocognitive testing; Other: MRI

INTERVENTIONS:
Radiation: Amyloid PET scan — Amyloid Positron Emission Tomography scan using radio tracer florbetapir-F18
Drug: Tau PET scan using MK-6240 — Tau Positron Emission Tomography scan using radio tracer MK-6240
  Other Names: tau PET
Behavioral: Neurocognitive testing — A battery of clinical neuropsychological assessments and computerized cognitive tasks will be used to test participants' memory and cognitive abilities.
Other: MRI — High-resolution structural, functional, and diffusion Magnetic Resonance Imaging scans will be collected during the study.

SUMMARY:
The purpose of this research study is to understand the factors that underlie changes in thinking and memory with increasing age. The investigators will test the usefulness of MRI, PET, and cognitive testing in detecting subtle changes in the brain that precede cognitive decline. An addendum to this study includes additional PET scans to examine the relationship between tau protein in the brain and cognitive decline. Tau is a protein that is known to form tangles in the areas of the brain important for memory, and these tau tangles are a hallmark of Alzheimer's disease. This sub-study research aims to look at the tau accumulation in the brain using an investigational drug called MK-6240, which is a radio tracer that gets injected prior to a positron emission tomography (PET) scan.

DETAILED DESCRIPTION:
This study investigates the relationship between Alzheimer's disease (AD) pathology, brain structure and function, as well as cognition in non-demented older adults. The goal is to develop a more complete understanding of the factors that lead to cognitive decline in the elderly and progression to AD. The investigators will enroll 200 cognitively intact adults between the ages of 60-85 years old from the UCI Alzheimer's Disease Research Center or directly from the local community. Study procedures will include: 1) PET amyloid scans with Amyvid™ radiotracer (florbetapir-F18) and PET tau scans with [18F]MK6240 radiotracer; 2) High-resolution structural, functional, and diffusion MRI; and 3) Cognitive examinations. The investigators will track cognitive outcomes through longitudinal monitoring. Amyloid imaging will only be conducted once in the study at baseline, and MRI and tau PET imaging will be at baseline and Year 1. The investigators aim to identify the best combination of tests for predicting longitudinal cognitive/clinical decline. The proposed study will significantly inform the understanding of cognitive decline in the aging brain and allow investigators to better define preclinical AD and make recommendations for future intervention trials.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 60 or older;
2. Speaks fluent English or Spanish;
3. Visual and auditory acuity adequate for neuropsychological and computerized testing;
4. Good general health with no disease(s) expected to interfere with the study;
5. Willing and able to participate for the duration of the study and in all study procedures including MRI and PET;
6. Normal cognition defined as a Clinical Dementia Rating of 0 and a Mini-Mental State Examination score of 25 or higher. FAST Stage 1 or 2.
7. Subjective memory or other cognitive complaints will be included.

Exclusion Criteria:

1. Significant co-morbid neurologic disease such as Parkinson's disease, multiple sclerosis, brain cyst, tumor or aneurysm;
2. Major health conditions, except for Type II diabetes mellitus, hypercholesterolemia, and hypertension, which are NOT exclusionary for this study given their high prevalence in our target populations;
3. Significant psychiatric disorders such as schizophrenia, bipolar disorder, or attention-deficit hyperactivity disorder, except for depression and anxiety, which are NOT exclusionary for this study given their high prevalence in our target populations;
4. Existing diagnosis of dementia or mild cognitive impairment;
5. Alcohol or substance abuse or dependence within the past 2 years (DSM-IV criteria);
6. MRI contraindications, e.g. pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments or foreign objects in the eyes, skin or body. Females who are pregnant or trying to get pregnant are also excluded;
7. PET contraindications, e.g. significant prior radiation exposure and pregnancy.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2026-12-22 (Estimated); Study Completion 2027-12-22 (Estimated)

PRIMARY OUTCOMES:
Change in Clinical Dementia Rating - Sum of Box Score | Years 4 and 5 of the grant
  A measure of cognitive/clinical decline

SECONDARY OUTCOMES:
Change in lure discrimination index - objects | Years 4 and 5 of the grant
  Key measure of performance on the object pattern separation task
Change in lure discrimination index - spatial | Years 4 and 5 of the grant
  Key measure of performance on the spatial pattern separation task
Change in lure discrimination index - temporal | Years 4 and 5 of the grant
  Key measure of performance on the temporal pattern separation task
Change in entorhinal cortical thickness | Years 4 and 5 of the grant
  Key measure of structural decline on MRI scans
Change in perforant path integrity | Years 4 and 5 of the grant
  Key measure of structural connectivity decline on MRI scans
Change in tau spatial distribution - advancing Braak stage | Years 4 and 5 of the grant
  Key measure of tau spatial spread on tau PET scans

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Yassa, PhD, Principal Investigator — University of California, Irvine; Liv C McMillan, BS, CCRP, Study Director — University of California, Irvine
Locations (1):
- University of California, Irvine, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stevenson RF, Reagh ZM, Chun AP, Murray EA, Yassa MA. Pattern Separation and Source Memory Engage Distinct Hippocampal and Neocortical Regions during Retrieval. J Neurosci. 2020 Jan 22;40(4):843-851. doi: 10.1523/JNEUROSCI.0564-19.2019. Epub 2019 Nov 20. PMID 31748377
- [Result] Holbrook AJ, Tustison NJ, Marquez F, Roberts J, Yassa MA, Gillen DL; Alzheimer's Disease Neuroimaging Initiative section sign. Anterolateral entorhinal cortex thickness as a new biomarker for early detection of Alzheimer's disease. Alzheimers Dement (Amst). 2020 Aug 25;12(1):e12068. doi: 10.1002/dad2.12068. eCollection 2020. PMID 32875052
- [Result] Chappel-Farley MG, Mander BA, Neikrug AB, Stehli A, Nan B, Grill JD, Yassa MA, Benca RM. Symptoms of obstructive sleep apnea are associated with less frequent exercise and worse subjective cognitive function across adulthood. Sleep. 2022 Mar 14;45(3):zsab240. doi: 10.1093/sleep/zsab240. PMID 34604910
- [Result] Adams JN, Kim S, Rizvi B, Sathishkumar M, Taylor L, Harris AL, Mikhail A, Keator DB, McMillan L, Yassa MA. Entorhinal-Hippocampal Circuit Integrity Is Related to Mnemonic Discrimination and Amyloid-beta Pathology in Older Adults. J Neurosci. 2022 Nov 16;42(46):8742-8753. doi: 10.1523/JNEUROSCI.1165-22.2022. Epub 2022 Oct 27. PMID 36302636
- [Result] Adams JN, Marquez F, Larson MS, Janecek JT, Miranda BA, Noche JA, Taylor L, Hollearn MK, McMillan L, Keator DB, Head E, Rissman RA, Yassa MA. Differential involvement of hippocampal subfields in the relationship between Alzheimer's pathology and memory interference in older adults. Alzheimers Dement (Amst). 2023 Apr 5;15(2):e12419. doi: 10.1002/dad2.12419. eCollection 2023 Apr-Jun. PMID 37035460
- See also: BEACoN (Biomarker Exploration in Aging, Cognition, and Neurodegeneration) study website — https://beacon.bio.uci.edu